CLINICAL TRIAL: NCT05556278
Title: Evaluation of Ecography as a Diagnostic Tool in the Carpal Tunnel Syndrome Compared to the Studies of Electroconduction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: RHB-02/2019
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; nerve conduction study; ultrasound; screening; diagnosis
MeSH Terms: conditions — Carpal Tunnel Syndrome; Disease | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: An electroneurography and an ultrasound study will be performed to patients with clinical suspicion of CTS and fulfilling the inclusion/exclusion criteria.
  Interventions: Diagnostic Test: Ultrasound study; Diagnostic Test: Neurophysiological test

INTERVENTIONS:
Diagnostic Test: Ultrasound study — based on the recommendations of the American Association of Electrodiagnostic Medicine (AAEM) (1)
Diagnostic Test: Neurophysiological test — ultrasound protocol described by Chen et al. (2)
  Other Names: Nerve conduction study

SUMMARY:
The main objective is to investigate the value of ultrasound in the diagnosis of Carpal Tunnel Syndrome (CTS), and among the secondary objectives, to establish the ultrasound parameters that are predictors of CTS in comparison with neurophysiological studies, attempting to standardize a protocol and reference values that determine the presence or absence of CTS. Finally, cost-effectiveness analysis is proposed.

DETAILED DESCRIPTION:
The reference test with which the ultrasound is compared is the neurophysiological test (NPT).

The expected timeline for the study is to be performed between July 2020 and May 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting clinical symptoms suggestive of CTS, at least one of the following:

   * Neuropathic profile pain in wrist-hand at the level of the median nerve territory (wrist, first-second-third, and radial half of the fourth finger by palmar and/or volar side), possibility of irradiation of the pain towards the forearm and/or arm.
   * Nocturnal symptoms.
   * Hypotrophy or atrophy of the thenar eminence.
   * Self-described sensory alteration (sensation of cramping, numbness, tingling, hypoalgesia or analgesia).
2. Age: 18 to 75 years.
3. Consent to participate in the study.

Exclusion Criteria:

1. Previous surgery on the wrist
2. Acquired or hereditary pathology causing peripheral neuropathies
3. Polyneuropathy of any etiology
4. Rheumatoid arthritis
5. Diabetes Mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of CTS that come consecutively from the Neurophysiology Department of the Virgen Macarena Hospital in Seville (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 438 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Demographic variables | January 2021 to September 2022
  Sex, age, time of evolution of the clinic, manual dominance, hand affected, body mass index, employment status, type of work (pink, white or blue collar), time worked, triggers of symptoms, what symptoms are relieved with, as well as toxic habits, whether they are smokers (to be answered affirmative or negative) or alcohol consumers (to be answered affirmative or negative).
Electrodiagnostic variables | January 2021 to September 2022
  Motor conduction velocity of the median nerve (calculating distal motor latency and wrist-elbow motor conduction velocity), motor conduction velocity of the ulnar nerve (calculating distal motor latency, lower and upper wrist-elbow motor conduction velocity), orthodromic sensory conduction of the median, ulnar and radial nerve, as well as antidromic sensory conduction of the median, ulnar and radial nerve.
Ultrasound variables | January 2021 to September 2022
  The cross-sectional area (CSA), range of median nerve thinning, wrist-forearm index, flexor retinaculum bulge, power Doppler uptake, and existence of notches
Boston Carpal Tunnel Questionnaire | January 2021 to September 2022
Cost evaluation | From September 2022 to May 2023
  Costs of the consumables established by the Andalusian Health Service used in both tests and the average time for each of the tests

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de la Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol can be accessed by contacting the trial team at (e-mail). Anonymized participants level data and statistical codes used for the analysis are available on request and subject to data sharing agreements. Data sharing may only be possible after relevant embedded trials have been published.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] American Association of Electrodiagnostic Medicine, American Academy of Neurology, and American Academy of Physical Medicine and Rehabilitation. Practice parameter for electrodiagnostic studies in carpal tunnel syndrome: summary statement. Muscle Nerve. 2002 Jun;25(6):918-22. doi: 10.1002/mus.10185. No abstract available. PMID 12115985
- [Background] Chen YT, Williams L, Zak MJ, Fredericson M. Review of Ultrasonography in the Diagnosis of Carpal Tunnel Syndrome and a Proposed Scanning Protocol. J Ultrasound Med. 2016 Nov;35(11):2311-2324. doi: 10.7863/ultra.15.12014. Epub 2016 Sep 14. PMID 27629754
- [Derived] Murciano Casas MP, Rodriguez-Pinero M, Jimenez Sarmiento AS, Alvarez Lopez M, Jimenez Jurado G. Evaluation of ultrasound as diagnostic tool in patients with clinical features suggestive of carpal tunnel syndrome in comparison to nerve conduction studies: Study protocol for a diagnostic testing study. PLoS One. 2023 Nov 10;18(11):e0281221. doi: 10.1371/journal.pone.0281221. eCollection 2023. PMID 37948425